CLINICAL TRIAL: NCT06926894
Title: Single Center Phase I Study of Adoptive Immunotherapy of Refractory Viral Infection With ex Vivo Expanded Rapidly Generated Virus Specific T (R-MVST) Cells for Immunodeficient Children and Young Adults
Brief Title: R-MVST Cells for Treatment of Viral Infections in Children and Young Adults
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Prakash Satwani, Professor of Pediatrics, Columbia University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AAAV1433
Record Dates: First submitted 2025-04-08; First posted 2025-04-15 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Epstein-Barr Virus; Cytomegalovirus Infections; Adenovirus; BK Virus Infection; Immune Deficiency
MeSH Terms: conditions — Epstein-Barr Virus Infections; Cytomegalovirus Infections; Adenoviridae Infections; Immunologic Deficiency Syndromes | interventions — Cell Count

STUDY DESIGN:
Intervention Model Description: Dose escalations will be performed separately for each group and will employ a classic 3+3 algorithmic design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A: Allogenic Stem Cell Transplant Recipients (Experimental): Patients who have infection due to cytomegalovirus (CMV), Epstein-Barr virus (EBV), adenovirus or BK virus, and are recipients of hematopoietic stem cell transplant.
  Interventions: Drug: Rapidly generated virus specific T (R-MVST) cells
- Group B: Solid Organ Transplant Recipients (Experimental): Patients who have infection due to cytomegalovirus (CMV), Epstein-Barr virus (EBV), adenovirus or BK virus, and are recipients of solid organ transplant.
  Interventions: Drug: Rapidly generated virus specific T (R-MVST) cells
- Group C: Other Immunocompromised Patients (Experimental): Patients who have infection due to cytomegalovirus (CMV), Epstein-Barr virus (EBV), adenovirus or BK virus, and are immunocompromised for reasons other than hematopoietic stem cell transplant or solid organ transplant.
  Interventions: Drug: Rapidly generated virus specific T (R-MVST) cells

INTERVENTIONS:
Drug: Rapidly generated virus specific T (R-MVST) cells — Group A dose escalation schedule:
  * Cohort (-1A): 0.25x10^6 R-MVST TNC/kg
  * Cohort (1A): 0.5x10^6 R-MVST TNC/kg
  * Cohort (2A): 1x10^6 R-MVST TNC/kg
  Groups B & C dose escalation schedule:
  * Cohort (-1B) + (-1C): 1x10^6 R-MVST TNC/kg
  * Cohort (1B) + (1C): 2x10^6 R-MVST TNC/kg
  * Cohort (2B) + (2C): 4x10^6 R-MVST TNC/kg
  Other Names: R-MVST infusion; total nucleated cells (TNC)

SUMMARY:
The primary objective is to determine the safety and feasibility of administering R-MVST cells to patients with refractory viral reactivation and/or symptomatic disease caused by Epstein Barr Virus (EBV), cytomegalovirus (CMV), adenovirus (ADV) or BK virus. R-MVST cells will be generated on-demand from the closest partially human leukocyte antigen (HLA)-matched (minimum haploidentical) healthy donors or from the original allo-transplant donor if available. The investigator will closely monitor the recipients for potential toxicities including graft-versus-host disease (GVHD) post-infusion.

Secondary objectives are to determine the effect of R-MVST infusion on viral load, possible recovery of antiviral immunity post-infusion and for evidence of clinical responses and overall survival. Recipients will be monitored for secondary graft failure at day 28 post R-MVST infusion.

DETAILED DESCRIPTION:
Starting from childhood, majority of healthy humans are exposed to common viruses such as CMV, EBV, BK and related human polyomaviruses and herpes viruses. Under normal circumstances those infections are well controlled by the adaptive immune system, but never eliminated. Instead, they are fairly inactive and produce relatively few consequences or symptoms. However, when T cell mediated immunity is suppressed, those dormant viruses reactivate and can cause a significant end-organ or severe systemic syndrome. This viral reactivation contributes to morbidity and mortality in recipients of allogeneic stem cell transplant (HCT) and solid organ transplants (SOT), and can affect many other patients who receive immunosuppressive therapies or have underlying pathology that affects T cell function, including patients with autoimmune diseases, congenital immunodeficiencies or HIV/AIDS. As a result of a weakened immune response, conventional antiviral prophylaxis or treatment with acyclovir and ganciclovir/foscarnet (for CMV) or rituximab (against EBV) are not always effective.

The main purpose of this study is to test whether giving an experimental cell product can treat the viral infection in patients who have conditions that cause poor function of their immune system, such as infections caused by viruses such as Cytomegalovirus (CMV), Epstein-Barr Virus (EBV), BK virus, or adenovirus. The cell product is called rapidly generated virus specific T cells or R-MVST.

This is a single center, Phase 1, non-randomized open-label dose escalation study in three groups of immunocompromised patients. The recipients of allogeneic HCT who will be enrolled in Group A, while SOT recipients will be enrolled in Group B and non-transplanted immunocompromised recipients will be enrolled in Group C. Each group will undergo independent dose escalation.

ELIGIBILITY:
Inclusion Criteria:

* Children and young adults (3 months to <26 years) of all ethnic groups will be eligible for the treatment
* Patients with history of HCT or SOT who demonstrate evidence of viral reactivation and/or infection manifesting as end-organ or systemic disease due to one or more of the following viruses: EBV, CMV, ADV or BK virus and suboptimal response to the standard of care therapy.
* Recurrent or Multiple Viral Infection. RVI defined as occurrence of more than one episode of reactivation that required intervention or symptomatic disease in recipient of allogeneic HCT that required standard of care treatment. MVI defined as more than one virus reactivating (defined by PCR positivity) or causing symptomatic systemic or end-organ disease. At least one of those viral reactivations required standard of care intervention. No standard of care therapy is defined for ADV and BK. Patients with multiple infections/reactivations will be eligible as long as at least one of those viral infections meet the criterium of "refractory".

Exclusion Criteria:

* Patients with other uncontrolled infections, except for CMV, EBV, ADV or BK. For bacterial infections, patients must be receiving definitive therapy and have no signs of progressing infection for 72 hours prior to the day of infusion. For fungal infections, patients must be receiving definitive systemic anti-fungal therapy and have no signs of progressing infection for 1 week prior to R-MVST infusion. Progressing infection is defined as hemodynamic instability attributable to sepsis or new symptoms, worsening physical signs or radiographic findings attributable to infection. Persisting fever without other signs or symptoms will not be interpreted as progressing infection.
* Patients who receive corticosteroids at ≥ 0.5mg/kg prednisone or equivalent.
* Patients who received anti-thymocyte globulin (ATG, Alemtuzumab (Campath), or other T-Cell immunosuppressive monoclonal antibodies in the last 28 days.
* Patients who received methotrexate, or other antimetabolite-type immunosuppressants that are toxic to proliferating T cells in the last 7 days.
* Patients who received extracorporeal photopheresis within the last 28 days.
* Patients who received checkpoint inhibitor agents (e.g., nivolumab, pembrolizumab, ipilimumab) within 3 drug half-lives of the most recent dose to the infusion of R-MVST.
* Received donor lymphocyte infusion in last 28 days.
* Evidence of GVHD ≥ grade 2
* Evidence of biopsy-proven acute rejection in SOT recipients
* Active and uncontrolled relapse of malignancy
* Patients who are pregnant, or breastfeeding.
* Female of childbearing potential, or male with a female partner of childbearing potential, unwilling to use a highly effective method of contraception.
* Uncontrolled intercurrent illness including, but not limited to symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients who have received investigational (IND) product within 14 days of infusion of the the R-MVST cells.
* Unable or unwilling to receive infusions at Morgan Stanley Children's Hospital.

Ages: 3 Months to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-04-20 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of toxicity that leads to safety endpoint | Up to 28 days post R-MVST infusion
  This is to measure the incidence of toxicity post-infusion. Toxicities to consider include: GI toxicity, renal toxicity, hemorrhagic toxicity, cardiovascular toxicity hypotension, cardiac arrhythmia and left ventricular systolic dysfunction), neurological toxicity (somnolence and seizure), coagulation toxicity, vascular toxicity and pulmonary toxicity.
Incidence of GVHD post-infusion that leads to safety endpoint | Up to 28 days post R-MVST infusion
  This is to measure the incidence of GVHD post-infusion. The safety endpoint will be defined as de novo acute GVHD grade IV within 28 days of the last dose of R-MVST, or grades 3-5 infusion related adverse events within 28 days of the last cytotoxic T-lymphocyte (CTL) dose, or grades 4-5 non-hematological adverse events within 28 days of the last CTL dose that are not due to the pre-existing infection or the original malignancy or pre-existing co-morbidities as defined by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0.

SECONDARY OUTCOMES:
Percentage of subjects with good response in viral load or end-organ disease improvement | Up to 1 year after the initial R-MVST infusion
  This is to measure the effect of R-MVST infusion on viral load and possible recovery of antiviral immunity post-infusion. Subjects with complete response, partial response and stable disease will be tallied.
  If patient has end-organ involvement, the disease will be monitored for the evidence of clinical response. In case of post-transplant lymphoproliferative disorder (PTLD)/EBV lymphoma, the standard Cheson criteria will be applied for adult patients.
Overall survival rate | Up to 1 year after the initial R-MVST infusion
  This is to measure the effect of R-MVST infusion on viral load and possible recovery of antiviral immunity post-infusion. The overall survival rate is defined as the percentage of people in a study or treatment group who are still alive for a certain period of time after they were diagnosed with or started treatment for a disease, such as cancer.
Incidence of secondary graft failure | Day 28 post R-MVST infusion
  Secondary graft failure is defined as initial neutrophil engraftment followed by subsequent decline in the absolute neutrophil count (ANC) to < 500/mm3 for three consecutive measurements on different days, unresponsive to growth factor therapy that persists for at least 14 days in the absence of a known cause such as relapse. Secondary graft failure will be assessed at 28 days post R-MVST infusion in allo-HCT recipients and in recipients of solid organ transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Prakash Satwani, MD, Principal Investigator — Professor of Pediatrics
Locations (1):
- Columbia University Medical Center / New-York Presbyterian, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No